CLINICAL TRIAL: NCT06370936
Title: The EXPLAIN Study: Exploring Plant-Based Meat Analogues for Their Impact on Health
Acronym: EXPLAIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Responsible Party: Principal Investigator, Lydia A. Afman, Associate professor, Wageningen University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: NL84824.091.23; NL84824.091.23 (Other: CCMO / Toetsingonline)
Record Dates: First submitted 2024-01-19; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Blood Pressure; Cardiometabolic Health
Keywords: Standardized diet; Plant based meat analogues; Blood pressure; Cardiometabolic health; Intestinal health; Microbiome; Animal meat

STUDY DESIGN:
Intervention Model Description: Participants will follow both an 8-week completely controlled dietary intervention followed by a 10-week washout period followed by another 8-week completely controlled dietary intervention.
Who Masked: Investigator
Masking Description: Treatment order (PBMA intervention - Meat intervention versus Meat intervention - PBMA intervention) is masked for the researchers. The order is not masked for participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Animal meats then PBMAs (Experimental): For the first treatment period of 8 weeks, participants receive a standardized diet with a variety of meat products, after a 10-week washout period this is followed by a standardized diet with a variety of PBMAs for the second treatment period.
  Interventions: Other: Standardized diet with commercially available animal meats (comparator products); Other: Standardized diet with commercially available PBMAs (intervention products)
- PBMAs then Animal meats (Experimental): For the first treatment period of 8 weeks, participants receive a standardized diet with a variety of PBMAs, after a 10-week washout period this is followed by a standardized diet with a variety of meat products for the second treatment period.
  Interventions: Other: Standardized diet with commercially available animal meats (comparator products); Other: Standardized diet with commercially available PBMAs (intervention products)

INTERVENTIONS:
Other: Standardized diet with commercially available animal meats (comparator products) — Fully controlled standardized diet with commercially available meats from animal origin. Fully controlled means that all food products 8-week intervention will be provided by the HNRU at Wageningen University. The standardized diet is designed to maintain body weight, and follows the average nutritional pattern of middle-aged men and women in the Netherlands, while taking individual habitual energy intake into account. The diet will have the same dietary composition for each person and energy intake will be based on the energy requirements of an individual. The diet is the same for both intervention periods, except for the origin of meat products: PBMAs versus meat of animal origin.
Other: Standardized diet with commercially available PBMAs (intervention products) — Fully controlled standardized diet with commercially available Plant-Based Meat Analogues (PBMAs). Fully controlled means that all food products 8-week intervention will be provided by the HNRU at Wageningen University. The standardized diet is designed to maintain body weight, and follows the average nutritional pattern of middle-aged men and women in the Netherlands, while taking individual habitual energy intake into account. The diet will have the same dietary composition for each person and energy intake will be based on the energy requirements of an individual. The diet is the same for both intervention periods, except for the origin of meat products: PBMAs versus meat of animal origin.

SUMMARY:
Plant-based diets with little to no meat are considered healthy and sustainable by the general public. The increasingly popular plant-based meat analogues (PBMAs) allow consumers to easily decrease meat intake while maintaining their dietary patterns. However, scientific knowledge on the health impact of PBMAs on humans is currently very limited.

The primary objective of this clinical trial is to evaluate if and to what extent replacing all meat products in an average Dutch diet with currently commercially available PBMAs affects the systolic blood pressure of middle-aged men and women in a 2x8 week fully dietary controlled crossover intervention study. The secondary objectives are to assess the effect of this replacement of meat products with PBMAs on cardiometabolic health, gut microbiome, intestinal health, well-being, and underlying biological mechanisms.

114 men and women with a BMI of 23-40 kg/m2, aged 45-75 years will be included in the study. Participants will follow both an 8-week completely controlled diet in which all meats are of plant-based origin (PBMAs) and an 8-week diet in which all meats are of animal origin in randomized order with a 10-week wash-out period. Before the intervention starts, the participants will be characterized to describe them on anthropometrics, glucose tolerance and insulin sensitivity, genetics, sleep patterns, and stress levels. Before the start and at the end of each 8-week dietary intervention period, several measurements, including systolic blood pressure monitoring and secondary outcome measures will be done. Additionally, systolic and diastolic blood pressure will be monitored throughout the dietary interventions and a small quantity of parameters related to the secondary objectives will be measured.

DETAILED DESCRIPTION:
Plant-based diets with little to no meat are considered healthy and sustainable by the general public. The increasingly popular plant-based meat analogues (PBMAs) allow consumers to easily decrease meat intake while maintaining their dietary patterns. PBMAs are designed to mimic the sensory and textural properties of meat and to replace animal protein with plant protein. Processing of plant-based ingredients is needed to achieve this, which potentially compromises the sustainability and health assets of PBMAs. One of the concerns with processing is that it results in relatively high salt levels in the products, which could affect the blood pressure of consumers. However, scientific knowledge on the health impact of PBMAs on humans is currently very limited. Therefore, a fully controlled dietary intervention with a standardized diet is needed to evaluate the health impact of commercially available PBMAs.

The primary objective is to evaluate if and to what extent replacing all meat products in an average Dutch diet with currently commercially available PBMAs affects the systolic blood pressure of middle-aged men and women in a 2x8 week fully dietary controlled crossover intervention study. The secondary objectives are to assess the effect of this replacement of meat products with PBMAs on cardiometabolic health, gut microbiome, and intestinal health, well-being, and underlying biological mechanisms. In addition, the investigators aim to study the relation between diet-specific responses (comparing PBMAs and meat products) and phenotype, including glucose responses and body composition.

The study compromises a randomized crossover fully controlled dietary intervention at Wageningen University which consists of 2x8 week interventions separated by a 10-week washout period. Before the intervention starts, the participants will be characterized to describe them on anthropometrics, glucose tolerance and insulin sensitivity, genetics, sleep patterns, and stress levels. Before the start and at the end of each 8-week dietary intervention period, several measurements, including systolic blood pressure monitoring and secondary outcome measures will be done. Additionally, systolic and diastolic blood pressure will be monitored throughout the dietary interventions and a small quantity of parameters related to the secondary objectives will be measured.

The study population consists of 114 men and women with a BMI of 23-40 kg/m2, aged 45-75 years, and weight stable (± <3kg) for at least three months before inclusion. Participants will follow both an 8-week completely controlled diet in which all meats are of plant-based origin (PBMAs) and an 8-week diet in which all meats are of animal origin in randomized order with a 10-week wash-out period. Diets are fully controlled which implies that all foods and meals are provided to participants by the Human Nutrition Research Unit (HNRU) and are based on participants' habitual energy needs to maintain a stable body weight throughout the study. Except for PBMAs/meat, all other foods will be identical in both intervention diets. The composition of the diets is based on the Dutch National Food Consumption Survey. All food products provided, including the PBMAs, are commercially available.

The total study duration for a participant will be a little over >6 months, including the 10-week washout. The total time that needs to be invested by participants in this study with visits and at-home measurements is 72 hours. Participants are restricted for a total of 16 weeks in their eating habits since they need to follow a fully standardized diet. Subjects will have their blood pressure measured at the HNRU and additionally will have to measure their blood pressure at home. In addition, subjects have to wear continuous glucose and physical activity monitors twice during the study for a total of approximately 28 days. During the characterization period, participants will visit the HNRU once or twice depending on participant preference. For the measurements before and at the end of each dietary intervention period, participants visit the HNRU three times per intervention period (one extra visit after for the HFMM), so six times total. Additionally, during the dietary intervention, participants will visit the Human Research Unit twice a week during dinner time.

ELIGIBILITY:
Inclusion Criteria:

* BMI of 23-40 kg/m2
* Age 45-75 years
* Willing to consume both meat and PBMAs
* Stable body weight (lost/gained ± <3 kg over the last 3 months prior to inclusion)

Exclusion Criteria:

* Diseases or prior surgeries affecting the stomach, liver, kidneys or intestines (allowed i.e. appendectomy)
* Food allergies, intolerances (including lactose/gluten intolerance) for products used in the study design, and/or dietary restrictions interfering with the study (including special diets, vegetarians, and eating disorders)
* Cardiovascular diseases (e.g. heart failure. But hypertension up to 160 mmHg is allowed for inclusion as indicated by the research physician) or cancer (e.g. non-invasive skin cancer allowed)
* Anemia defined as Hb concentrations <8.5 mmol/L for men and <7.5 mmol/L for women
* Diagnosed with type 1 or type 2 diabetes
* Blood pressure >160 mmHg*
* Major mental disorders
* Drug-treated thyroid diseases (well-substituted hypothyroidism is allowed for inclusion)
* Diseases with a life expectation shorter than 5 years
* Regular use of/receiving medication interfering with research outcomes (as judged by research physician), such as the use of glucose-lowering drugs, insulin, use of medication that impacts gastric emptying, use of antipsychotics
* Starting or changing blood pressure medication type or dose during the study. (Continuation of blood pressure medication usage is allowed during the study)
* Use of anti-biotics over the last 3 months before the study start
* Dietary habits interfering with study design (vegan/vegetarian, ketogenic diet, etc.)
* Intention to change the intensity of exercise during the study period;
* Intention to lose weight during the study period
* Current smokers (including use of e-cigarettes)
* Use of soft and/or hard drugs (cannabis included)
* Abuse of alcohol (alcohol consumption defined as >14 glasses (women) or >21 glasses (men) of alcoholic beverages per week)
* Use of strong vitamins or other dietary supplements (e.g. iron- or B12-supplements, pre- or probiotics) expected to interfere with the study outcomes.
* Donated blood within 2 months prior to the screening
* Inability to comply with the study diet
* Being pregnant or lactating or planning to become pregnant
* Unable/unwilling to download a research application on the mobile phone
* Inability to understand study information and/or communicate with staff
* Inability/unwillingness to comply with staff instructions
* Displaying misbehavior towards other participants/staff
* Participation in another study that involves an intervention within two months prior to the intervention
* Working or doing a thesis/internship at the Division of Human Nutrition and Health or the Laboratory of Microbiology of Wageningen University.

[*Participants with a screening systolic blood pressure >140 mmHg - ≤160 mmHg need written permission for participation without having (medical) treatment for the study period granted by their general practitioner after assessment of their cardiovascular risk. Participants within this screening range who cannot hand over written clearance from their general practitioner will be excluded from participation. Participants whose blood pressure has measured >140 mmHg (systolic) or >90 mmHg (diastolic) one or more times during the study, will receive a letter for referral to the general practitioner.]

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Systolic blood pressure | 12 times during the trial, 6 times per 8-week intervention (1 time before intervention period, then biweekly measurements, and 1 measurements in week 8 of 8-week intervention)
  Systolic blood pressure as measured with in-clinic blood pressure measurements

SECONDARY OUTCOMES:
Diastolic blood pressure | 12 times during the trial, 6 times per 8-week intervention (1 time before intervention period, then biweekly measurements, and 1 measurements in week 8 of 8-week intervention)
  Diastolic blood pressure as measured with in-clinic blood pressure measurements
Home systolic blood pressure | Twice daily for 16 weeks total (both 8-week interventions)
  Systolic blood pressure as measured by participant at-home
Home diastolic blood pressure | Twice daily for 16 weeks total (both 8-week interventions)
  Diastolic blood pressure as measured by participant at-home
Home heart rate | Twice daily for 16 weeks total (both 8-week interventions)
  Heart rate as measured by participant at-home with blood pressure monitor
Fasting blood HbA1c levels | 4 times during the trial. 2 times per 8 week-intervention (1 time before intervention and 1 time during week 8 of 8-week intervention)
  Fasting HbA1c concentration
Fasting blood glucose levels | 4 times during the trial. 2 times per 8 week-intervention (1 time before intervention and 1 time during week 8 of 8-week intervention)
  Fasting glucose concentration
Fasting blood insulin levels | 4 times during the trial. 2 times per 8 week-intervention (1 time before intervention and 1 time during week 8 of 8-week intervention)
  Fasting insulin concentration
Fasting blood lipid spectrum | 4 times during the trial. 2 times per 8 week-intervention (1 time before intervention and 1 time during week 8 of 8-week intervention)
  Metabolomic analysis to determine all circulating blood lipids, including all cholesterol types, triglycerides and free fatty acids
Fasting blood metabolite profile | 4 times during the trial. 2 times per 8 week-intervention (1 time before intervention and 1 time during week 8 of 8-week intervention)
  Fasting blood metabolome as determined by metabolomics.
Fasting blood proteomic profile | 4 times during the trial. 2 times per 8 week-intervention (1 time before intervention and 1 time during week 8 of 8-week intervention)
  Proteomic analysis of fasting blood, incorporating an O-link panel, to determine circulating blood proteins, including protein biomarkers for inflammation such as cytokines.
Fasting blood cell transcriptomic profile | 4 times during the trial. 2 times per 8 week-intervention (1 time before intervention and 1 time during week 8 of 8-week intervention)
  Analysis of blood cells using transcriptomics to determine the blood transcriptome.
Fasting blood nutritional status | 4 times during the trial. 2 times per 8 week-intervention (1 time before intervention and 1 time during week 8 of 8-week intervention)
  Circulating vitamins and minerals related to meat and plant-based meat intake, including important circulating vitamins such as vitamins B6, B12, and D, and minerals such as markers of iron status, zinc, magnesium, and calcium.
Blood immune markers | 4 times during the trial. 2 times per 8 week-intervention (1 time before intervention and 1 time during week 8 of 8-week intervention)
  Blood immune- and immune-metabolism markers. This includes immune-related proteins including cytokines.
Blood immune cell populations | 4 times during the trial. 2 times per 8 week-intervention (1 time before intervention and 1 time during week 8 of 8-week intervention)
  Blood (immune) cell subpopulations. This compromises of whole blood CD45+ cell subset abundance such as abundance of T-lymphocytes and B-lymphocytes.
Metabolites in 24-hour urine | 4 times during the trial. 2 times per 8 week-intervention (1 time before intervention and 1 time during week 8 of 8-week intervention)
  Metabolomic analysis of urine collected over 24 hours, including markers for sodium excretion, urea nitrogen excretion, kidney function and consumption of (plant-based) meat, pH, and volume of urine.
Interstitial glucose profile | 4 weeks during trial, 2 continuous weeks per 8-week intervention
  Interstitial glucose concentrations, as measured by continuous glucose monitoring.
Physical activity | 4 weeks during trial, 2 continuous weeks per 8-week intervention
  Continuous physical activity levels, measured by the Actigraph accelerometer wGT3X-BT (ActiGraph, Pensacola, USA)
Fecal microbiome composition | 18 times during trial. Done 1 time before each 8-week intervention and weekly during 8-week intervention.
  Microbiome composition in the feces.
Fasting and postprandial circulating metabolites with a high fat mixed meal (HFMM) challenge | 2 times during the trial. 1 time at the end of each 8 week-intervention.
  Circulating fasting and postprandial metabolites upon a high-fat mixed meal (HFMM). At t=0, 30, 60, 90, 120, 180, and 240 minutes after the consumption of the HFMM blood is collected. This measurement is only for participants with veins suitable for a Venflon catheter.
Oral microbiome composition | 4 times during the trial. 2 times per 8 week-intervention (1 time before intervention and 1 time during week 8 of 8-week intervention)
  Microbiome composition in saliva.
Microbiome metabolites | 18 times during trial. Done 1 time before each 8-week intervention and weekly during 8-week intervention.
  Microbial metabolites of interest, such as SCFAs will be measured using high-performance liquid chromatography (HPLC).
Microbiome functionality | 18 times during trial. Done 1 time before each 8-week intervention and weekly during 8-week intervention.
  Microbiome functionality and genetic composition is assessed using batch-fermentation.
Self-reported gastro-intestinal symptoms | 18 times during trial. Done 1 time before each 8-week intervention and weekly during 8-week intervention.
  Gastro-intestinal symptoms as measured using the GSRS questionnaire (gastro-intestinal rating scale). The GSRS contains five scales: reflux syndrome, abdominal pain, constipation syndrome, diarrhoea syndrome and indigestion syndrome. Scores between 1-7. Low scores indicated absence or mild presence of symptoms, high scores indicated heavy presence of symptoms.
Self-reported constipation | 18 times during trial. Done 1 time before each 8-week intervention and weekly during 8-week intervention.
  Gastro-intestinal obstipation symptoms as measured using the PAC-SYM questionnaire (Patient Assessment of Constipation Symptoms). Scores between 1-4. Low scores indicated absence or mild presence of symptoms, high scores indicated heavy presence of symptoms.
Self-reported stool consistency and frequency | 18 times during trial. Done 1 time before each 8-week intervention and weekly during 8-week intervention.
  Self-reported stool consistency and frequency by using the Bristol Stool Chart (BSC) (scores between 1-7). Low scores indicate constipation and high scores diarrhea. Scores of 3-4 indicate a 'normal' stool.
Gastro-intestinal transit time | 4 times during the trial. 2 times per 8 week-intervention (1 time before intervention and 1 time during week 8 of 8-week intervention)
  Transit time measured using the blue dye method
Self reported product-specific attitude towards meat and PBMAs | 6 times during trial. 3 times per 8-week intervention, during CGM (continuous glucose monitor) wearing period.
  Self-reported product-specific attitude towards meat and PBMAs as measured using a questionnaire. Scores between 1-7. Low scores indicate a negative attitude toward the product, and high scores indicate a positive attitude toward the product.
Self reported meal-specific satiety with meat and PBMAs | 6 times during trial. 3 times per 8-week intervention, during CGM (continuous glucose monitor) wearing period.
  Self reported meal-specific satiety with meat and PBMAs measured using a questionnaire. The Visual Analogue Scale (VAS) is used for questions about satiety and Likert scale is used to assess the intensity of product attributes. Low scores indicate low liking/experience, and high scores indicate high liking/experience.
Self-reported general attitude toward meat and PBMAs | 10 times during trial. 5 times per 8-week intervention (before intervention, week 1,2,4 and 8).
  Self-reported general attitude toward meat and PBMAs as measured using a questionnaire. Scores between 1-7. Low scores indicate a negative general attitude and high scores indicate a positive general attitude

OTHER OUTCOMES:
Body composition | Baseline
  Body composition as measured by DEXA (Dual Energy X-ray Absorptiometry).
Genetic variation | Baseline
  Single Nucleotide Polymorphisms (SNPs) in genes relevant for metabolism and responses to food, collected using a mouth swab and/or buffycoat.
Oral glucose tolerance test (OGTT) | Baseline
  A 6-point OGTT measuring fasting and postprandial glucose and insulin responses. At t=0, 15, 30, 45, 60, 90, and 120 minutes, blood will be collected to measure plasma glucose and insulin concentrations. At t=0, HbA1c concentrations will also be determined. This measurement is only for participants with veins suitable for a Venflon catheter.
Habitual dietary intake | Baseline
  Habitual dietary intake assessment with a food frequency questionnaire (FFQ).
Perceived stress | Baseline
  Perceived stress of participant over past month as measured with the Perceived Stress Scale (PSS-10)
Chronotype assessment | Baseline
  Chronotype assessment of participant with reduced Morning-Eveningness Questionnaire (rMEQ)
Sleeping habits | Baseline
  Sleeping habits of participants over the past month as measured using the Pittsburgh Sleep Quality Index (PSQI).
Self reported habitual meat and PBMA consumption | 3 times during trial. At baseline and 2 times during 10-week washout period.
  Habitual dietary meat and PBMA consumption assessment using a questionnaire.
24-hour dietary recall | 6 times during the 10-week washout period
  24-hour dietary recall done using the Traqq mobile phone application.
Home environment microbiome composition | 4 times during the trial. 2 times per 8 week-intervention (1 time before intervention and 1 time during week 8 of 8-week intervention)
  Microbiome composition on electrostatic dust collectors (EDC) that are placed in participants home for 2 consecutive weeks accompanied with regarding geographic location and placement of EDC.

CONTACTS AND LOCATIONS:
Overall Officials: Lydia Afman, Principal Investigator — Wageningen University and Research
Locations (1):
- Wageningen University, Division of Human Nutrition, Wageningen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No